CLINICAL TRIAL: NCT04991272
Title: Effect of 10 Minutes Prewarming and Warmed Intravenous Fluid on Core Temperature in Patients Undergoing Urologic Surgery Under General Anesthesia
Brief Title: 10 Minutes Prewarming and Warmed Intravenous Fluid on Core Temperature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, In-Jung Jun, MD. PhD. associate Professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-05-004
Record Dates: First submitted 2021-07-16; First posted 2021-08-05 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Urologic Diseases
Keywords: hypothermia
MeSH Terms: conditions — Urologic Diseases; Hypothermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- warming group (Active Comparator): Warming group patients are applied prewarming with bair-hugger (43'C)(warm touch, COVIDIEN, full body blanket) for 10 minutes in the preanesthetic unit prior to induction of anesthesia. During operation, prewarmed intravenous fluid which was stored in the warming cabinet for more than 8 hours is connected and infused. Forced air blanket (warm touch, COVIDIEN, upper body blanket) with 38'C is applied for all patients during the operation.
  Interventions: Other: prewarming and warmed fluid infusion
- no warming group (No Intervention): No warming group patients are not applied prewarming devices. Intravenous fluid stored in room air is connected and infused during the operation. Forced air blanket (warm touch, COVIDIEN, upper body blanket) with 38'C is applied for all patients during the operation.

INTERVENTIONS:
Other: prewarming and warmed fluid infusion — prewarming with forced air warming system and warmed fluid infusion.
  Arms: warming group

SUMMARY:
Hypothermia occurs frequently during general anesthesia. This study is to evaluate the efficacy of 10 minutes of prewarming and warmed fluid during urologic surgery.

DETAILED DESCRIPTION:
During general anesthesia, vasodilation distributes body heat and leads to hypothermia. Especially during urologic operation (transurethral resection of bladder and prostate), bladder irrigation worsens hypothermia. Hence, various methods are used to maintain core temperature during operation.

Previous studies have demonstrated that prewarming of the patient is effective in maintaining core temperature perioperatively. However, more than 50% of patients who have applied prewarming for more than 30 minutes preoperatively are reported to fall in hypothermia. Hence, developing simple and effective method to prevent hypothermia is expected.

Hence, the investigators planned to examine the effect of active warming (10 minutes of prewarming preoperatively and prewarmed intravenous fluid intraoperatively) on hypothermia in patients undergoing urologic operation under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing urologic surgery(transurethral resection of bladder, prostate)

Exclusion Criteria:

* moderate to severe cardiopulmonary, renal impairment
* thyroid disease
* any infection sign
* abnormal temperature prior to induction of general anesthesia (<36'C or >37.5'C)
* refusal to participate in the study
* unable to understand the study

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
incidence of hypothermia at the end of the operation | approximately 1-2hours after induction (at the end of operation)
  after completion of the operation, number of patients with hypothermia (<36'C) using esophageal stethoscope will be recorded.

SECONDARY OUTCOMES:
change in temperature before and end of operation | on arrival at the OR upto 1-2hours after induction (at the end of the operation)
  change in core temperature will be calculated and compared
incidence of shivering | upto 1 hour after end of the operation (on arrival at the postanesthesia care unit)
  shivering will be evaluated using 4 point shivering scale (0=none, 1=core and neck shivering, 2= upper extremity 3= whole body)
thermal comfort | upto 1hour after end of the operation (at discharge of postanesthesia care unit)
  thermal comfort will be evaluated using thermal comfort scale ( 0= very cold, 5= fine, 10= very hot and uncomfortable)

CONTACTS AND LOCATIONS:
Overall Officials: In-Jung Jun, MD. PhD, Principal Investigator — Associate professor
Locations (1):
- Sanggye Paik Hospital, Seoul, South Korea